CLINICAL TRIAL: NCT00614081
Title: Measurement of Glomerular Filtration Rate With Contrast-enhanced Dynamic MR Imaging in Renal Transplant Recipients: Evaluation of the Agreement With the Cr51 -EDTA Method and of Reproducibility
Brief Title: GFR Measurement With Contrast-enhanced Dynamic MRI
Acronym: IREN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 7825; 2005-029
Record Dates: First submitted 2007-11-22; First posted 2008-02-13 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Transplantation, Kidney; Graft Occlusion, Vascular
Keywords: Glomerular filtration rate measurement; Contrast-enhanced dynamic MR imaging; Renal transplant recipients
MeSH Terms: conditions — Graft Occlusion, Vascular | interventions — Dynamic Contrast Enhanced Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Renal transplant recipients
  Interventions: Device: Contrast-enhanced dynamic MRI

INTERVENTIONS:
Device: Contrast-enhanced dynamic MRI

SUMMARY:
The aim of the study is to optimize and validate this MR-based GFR measurement in patients with a renal transplant, compared with the reference method, the Cr51- EDTA method: to select the most accurate combination of post-treatment of renal MR images and then evaluate its intra- and inter-rater reliability.

DETAILED DESCRIPTION:
Cr51- EDTA method is considered the reference method for measurement of glomerular filtration rate (GFR). However, this method requires several hours and several blood and urinary samplings. Therefore, the ability to get access to this parameter with a simple, valid and reliable method would be a significant progress in clinical follow-up of patients with renal disease. Contrast-enhanced dynamic MRI is now able to give this access to functional parameters as GFR, rapidly and non invasively, becoming an alternative to Cr51-EDTA method. If the acquisition method has been optimized, some problems remain unsolved: is the movement correction worthwhile for the accuracy of the measurement ? Which model provides the most accurate results ? What is the best way to calculate the total GFR (addition of all the voxels or the product of a mean value by the cortical volume)? These questions can be answered only by a comparison with a reference method.

The reference method will be performed after standard hydration, with intravenous injection of 100 µCi of Cr51- EDTA and urinary and blood samplings every 30 minutes during 3h. Dynamic MRI will be performed with fast 3D T1-weighted gradient-echo sequences during 5 minutes after injection of a third of a clinical dose of gadolinium. Post-treatment of images will be done on an off-line program allowing movement correction, conversion of signal intensity into concentration and application of different models. 8 combinations of post-treatment will be tested and compared to the reference method.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a renal transplant presenting with a graft dysfunction or a suspicion of vascular complication (renal artery stenosis…) or of urinary complication (dilatation of excretory system, collection) justifying to perform a non urgent MR examination
* Calculated glomerular clearance (MDRD method) > 20 ml/min
* Age ≥ 18 yo at the time of inclusion
* Negative pregnancy test
* Affiliation to the Social Security
* Written informed consent signed

Exclusion Criteria:

* Contra-indication to MRI: neurovascular clips, pacemaker, cochlear implant, orbital metallic object, claustrophobic patients…
* Contra-indication to gadolinium: previous hypersensitivity to Gd-Chelates
* Pregnancy or breastfeeding women
* Adult under legal supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
GFR according to MRI and Cr51 measurements on the same day | The same day

CONTACTS AND LOCATIONS:
Overall Officials: PEREZ Paul, Dr, Study Chair — University Hospital, Bordeaux, France
Locations (1):
- Service d'imagerie Diagnostique et interventionelle de l'adulte, Hôpital Pellegrin, CHU de Bordeaux, Bordeaux, France